CLINICAL TRIAL: NCT06492941
Title: A Randomized, Double-blind, Multicenter Phase Ⅲ Clinical Study of Docetaxel for Injection (Albumin Bound) Combined With Best Supportive Care Versus Placebo Plus Best Supportive Care in Advanced Pancreatic Cancer
Brief Title: A Study of Docetaxel for Injection (Albumin Bound) in Patients With Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB1801-011
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — Docetaxel; Injections

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to Docetaxel for Injection (Albumin Bound ) in combination with best supportive care or placebo in combination with best supportive care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel for Injection (Albumin Bound) in combination with best supportive care (Experimental): Docetaxel for Injection (Albumin Bound) ：i.v., q3w,100mg/m^2； Best supportive care includes, but is not limited to, pain control, nutritional support, and psychological care
  Interventions: Drug: Docetaxel for Injection (Albumin bound); Drug: Best supportive care
- Placebo in combination with best supportive care (Placebo Comparator): Placebo ：i.v., q3w； Best supportive care includes, but is not limited to, pain control, nutritional support, and psychological care
  Interventions: Drug: Placebo; Drug: Best supportive care

INTERVENTIONS:
Drug: Docetaxel for Injection (Albumin bound) — Docetaxel for Injection (Albumin bound), by intravenous infusion, every 3 weeks.
  Arms: Docetaxel for Injection (Albumin Bound) in combination with best supportive care
Drug: Placebo — Placebo was human blood albumin without the active ingredient docetaxel
  Arms: Placebo in combination with best supportive care
Drug: Best supportive care — Best supportive care includes, but is not limited to, pain control, nutritional support, and psychological care.

SUMMARY:
This study is a randomized, double-blind, multicenter, phase Ⅲ clinical study to compare the clinical efficacy and safety of Docetaxel for Injection (Albumin Bound) in combination with best supportive care versus placebo in combination with best supportive care in participants with pancreatic cancer who have received gemcitabine-containing and fluorouracil-containing regimens.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multicenter, phase Ⅲ clinical study to compare the clinical efficacy and safety of Docetaxel for Injection (Albumin bound) plus best supportive care versus placebo plus best supportive care in participants with pancreatic cancer who have received a previous treatment regimen containing gemcitabine and fluorouracil. It is planned to enroll 142 participants, and participants will be randomized to receive Docetaxel for Injection (albumin bound) in combination with best supportive care or placebo in combination with best supportive care in a 2:1 ratio. Best supportive care includes, but is not limited to, pain control, nutritional support, and psychological care.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged ≥18 years (subject to the date when the informed consent form is signed) and voluntarily signed the informed consent form.
* 2. Histologically or cytologically confirmed diagnosis of pancreatic cancer (including adenosquamous carcinoma).
* 3. Patients who have got disease progression or toxic intolerance after previous standard treatment (gemcitabine based and fluorouracil based therapy).
* 4. At least one evaluable lesion according to RECIST 1.1 .
* 5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* 6. Patients with fine organ function (no medical supportive treatments such as blood component transfusion, growth factors within 2 weeks before taking the relevant inspections):

  1. ANC≥1.5×10^9/L；
  2. Hb≥90 g/L；
  3. PLT≥100×10^9/L；
  4. ALB≥30 g/L；
  5. CR≤1.5× ULN and creatinine clearance≥40 mL/min（Cockcroft-Gault）；
  6. Total bilirubin≤1.5 × ULN(≤ 2 × ULN for patients with obstructive jaundice, ≤3 × ULN for patients with Gilbert's syndrome)；
  7. ALT and AST ≤ 3× ULN (≤5× ULN for patients with liver metastasis)；
  8. ALP≤2.5× ULN；
  9. PT、INR≤1.5×ULN。
* 7. The patient must agree to take adequate contraception from signing of ICF through 6 months after last dose, women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

* 1. Patients who have a history of severe allergy to any excipients of the investigational drug or taxanes，or known allergy and/or contraindications to glucocorticoids (including but not limited to active digestive tract ulcers, severe hypertension, severe hypokalemia, glaucoma, etc.).
* 2. Patients with partial or complete intestinal obstruction or complete biliary obstruction that cannot be relieved by active treatment.
* 3. Previous history of inflammatory bowel disease, chronic diarrhea, and gastrointestinal bleeding.
* 4. Patients who had a history of other active malignant tumors within 2 years before the first dose of the investigational drug, except for the study disease pancreatic cancer and curable cancer that had been cured (such as basal cell or squamous cell skin cancer, superficial bladder cancer, cervical cancer or breast cancer in situ that had been excised).
* 5. Patients with active hepatitis B (HBsAg and/or HBcAb positive but HBV DNA < 2000 IU/mL can be included), active hepatitis C (HCV antibody positive but HCV RNA negative can be included), and HIV antibody positive.
* 6. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for alopecia, hyperpigmentation, or other toxicity without safety risk judged by the investigator).
* 7. Patients with a history of severe cardiovascular disease, including but not limited to:：

  1. Severe heart rhythm or conduction abnormalities, including but not limited to ventricular arrhythmia requiring clinical intervention and third degree atrioventricular block within 6 months before the first dose of the investigational drug；
  2. History of myocardial infarction, unstable angina pectoris, angioplasty and coronary artery bypass surgery within 6 months before the first dose of the investigational drug;；
  3. Heart failure with New York Heart Association (NYHA) Classification of Class Ш and above；
  4. Long QTc syndrome or QTc > 480 msec；
  5. Poorly controlled hypertension (Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening period).
* 8. Patients with uncontrolled serous cavity effusion requiring frequent drainage or medical intervention (e.g., pleural effusion, abdominal effusion, pericardial effusion, etc., additional intervention was needed within 2 weeks after intervention, excluding exfoliative cytology testing of the exudate) within 2 weeks before the first dose of the investigational drug.
* 9. Patients with severe or active infections (including tuberculous infections) that require systemic antibacterial, antifungal, or antiviral therapy within 14 days before the first dose of the investigational drug, antiviral therapy for patients with viral hepatitis is permitted.
* 10. Received any anti-tumor therapy (including chemotherapy, targeted therapy, immunotherapy, etc.) and any clinical trial intervention within 4 weeks prior to the first use of the investigational drug or within 5 half-lives of the most recently used anti-tumor drug (whichever is shorter), and used traditional Chinese medicine or proprietary Chinese medicine with anti-tumor indications within 14 days before the first use of the investigational drug.
* 11. Patients who have used potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of the investigational drug.
* 12. Patients who have undergone major surgery within 4 weeks before the first dose of the investigational drug and had not recovered sufficiently, or who need to undergo major surgery during the study.
* 13. Pregnant or nursing women.
* 14. Patients who is participating in another clinical study simultaneously unless it is an observational (non-interventional) clinical study or within the follow-up period of an interventional study.
* 15. Other situations that the investigator considers not suitable for participating in the clinical study, including but not limited to: the patient is complicated by severe or uncontrolled medical conditions, which will increase the safety risk, interfere with the interpretation of study results or affect the study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
OS | Up to approximately 2 years
  The overall survival (OS) of the two groups. All the participants received tumor assessment every 6 weeks according to RECIST1.1.

SECONDARY OUTCOMES:
PFS | Up to approximately 2 years
  All the participants received tumor assessment every 6 weeks according to RECIST1.1 to evaluate the progression-free survival (PFS) .
ORR | Up to approximately 2 years
  All the participants received tumor assessment every 6 weeks according to RECIST1.1 to evaluate the objective response rate (ORR).
DCR | Up to approximately 2 years
  All the participants received tumor assessment every 6 weeks according to RECIST1.1 to evaluate the disease control rate (DCR).
DOR | Up to approximately 2 years
  All the participants received tumor assessment every 6 weeks according to RECIST1.1 to evaluate the duration of response (DOR).
Incidence of AE and SAE | Up to approximately 2 years
  Incidence of AE and SAE
PK | At the end of Cycle 1(each cycle is 21 days)
  Plasma concentration of docetaxel (free and total)

IPD SHARING:
Plan to Share IPD: No